CLINICAL TRIAL: NCT02582034
Title: Selective Internal Radiation Therapy for Hepatocellular Carcinomas With Yttrium-90 Loaded Microspheres: Optimized Dosimetry Versus Standard Dosimetry
Brief Title: Internal Radiation Therapy for Hepatocellular Carcinomas With Therasphere: Optimized Dosimetry Versus Standard Dosimetry
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOSISPHERES-01
Record Dates: First submitted 2015-10-09; First posted 2015-10-21 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Adenoma, Liver Cell
Keywords: Optimized Dosimetry versus standard Dosimetry; Internal Radiation Therapy
MeSH Terms: conditions — Adenoma, Liver Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dosimetry (Active Comparator): Standard Internal Radiation Therapy : Dose of radiation delivered to the tumoral volume is fixed : 120 Gray (GY)
  Interventions: Radiation: Standard Internal Radiation Therapy
- Optimized dosimetry (Experimental): Optimized Internal Radiation Therapy : Dose of radiation absorbed by the tumor is > 205 GY, if possible 250 or 300 Gy.
  Interventions: Radiation: Optimized Internal Radiation Therapy

INTERVENTIONS:
Radiation: Optimized Internal Radiation Therapy — Injection of yttrium-90 microspheres (TheraSphere®) is performed during the therapeutic angiogram, directly into the hepatic artery (left or right, or even segmental).
  Optimized dosimetry arm: the activity to be administered is calculated so as to deliver predictive dosimetry:
  * An absorbed dose to the tumor of at least ≥ 205 Gy and if possible exceeding 250 Gy or even 300 Gy
  * A dose at the treated healthy liver < 120 Gy in case of lobar treatment
  * Dose to the treated healthy liver can exceed 120 Gy in case of segmental treatment and hepatic reserve > 30%
  * A pulmonary dose < 30 Gy for one treatment and < 50 Gy in cumulative dose in case of multiple treatments.
  Arms: Optimized dosimetry
Radiation: Standard Internal Radiation Therapy — Injection of yttrium-90 microspheres (TheraSphere®) is performed during the therapeutic angiogram, directly into the hepatic artery (left or right, or even segmental).Standard dosimetry arm: the activity to be administered is calculated so as predictive dosimetry:
  * An absorbed dose of 120 ± 20 Gy to the treated volume (whatever the tumor absorbed dose)
  * A pulmonary dose < 30 Gy for one treatment and < 50 Gy in cumulative dose in case of multiple treatments.
  Arms: Standard dosimetry

SUMMARY:
The purpose of this study is to determine whether a treatment with Therasphere which is optimized is more efficient compared to a standard treatment for patients suffering from hepatocellular carcinomas.

DETAILED DESCRIPTION:
For patients suffering from hepatocellular carcinoma, a palliative treatment can be proposed if tumor expansion is limited to the liver. One of palliative treatment is the the Selective Internal Radiation Therapy (SIRT) with Therasphere®. This treatment is made secure by performing a diagnostic angiogram coupled with a hepatic perfusion scintigraph with which patients at risk of complications are identified and excluded. The treatment objective, with the standard dosimetric approach, is to deliver an absorbed dose of 120 ± 20 Gy to the treated hepatic volume, most often one lobe. Recent retrospective trials show that an optimized dosimetric approach, considering the dose absorbed by the tumor, is technically achievable and would probably make it possible to obtain a better effectiveness. In our experience, treatment personalisation have been described to be used for 60% of the patients with a tumor larger than 7 cm underlying the clinical impact of this new approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18,
* Written free and informed consent,
* Histologically demonstrated Hepatocellular Carcinoma (HCC), not a candidate for surgery or local ablative treatment (radio frequency, etc.)
* Barcelona Clinic Liver Cancer (BCLC) classification A, B or C,
* At least one lesion ≥ 7 cm,
* Hepatic reserve (hepatic parenchyma not treated) after the first SIRT ≥ 30%,
* Unilateral involvement, minimal bilateral involvement allowed only with a hepatic reserve ≥ 30% after SIRT
* Child A classification only, or B but with bilirubinemia <35 micromol/L,
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1,
* Patients whose biological parameters meet the following criteria:

  * Hemoglobin ≥ 8.5 g/dL,
  * Granulocytes ≥ 1500/mm3,
  * Platelets ≥ 50,000/mm3,
  * Bilirubinemia <35 micromol per liter,
  * Transaminases ≤ five times the upper limit of normal,
  * Creatininemia ≤ 1.5 times the normal upper limit,
* Expected survival over 12 weeks,
* Negative pregnancy test for women of childbearing age,
* If sorafenib has been taken the diagnostic angiogram must follow it by at least four weeks after its stop.

Exclusion Criteria:

* HCC operable or accessible to a local ablative treatment (radio frequency),
* Hepatectomy history unless a segmental treatment is considered, with a hepatic reserve ≥ 30% after SIRT,
* Prior treatment with sorafenib unless stopped at least four weeks earlier,
* History of chemo-embolization of the principal lesion, except in case of nodular residual lesion measuring at least 7 cm or in case of progression after initial response,
* Bilateral disease requiring a whole liver injection or with a hepatic reserve < 30% after SIRT
* Treatment of another cancer less than one year earlier,
* Extra-hepatic metastases other than adenopathies of the hilum smaller than 2 cm,
* >70% tumor invasion of the liver,
* Bilirubinemia ≥ 35 µmol/L,
* A Severe underlying biliary pathology:
* Bile duct anomaly (stent, dilation) Cirrhosis of biliary origin,
* Women of childbearing age without contraception
* Pregnant or nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to compare the response rate of the treated lesion at the first radioembolization, evaluated using European Association for the Study of the Liver (EASL) criteria of yttrium-90 marked glass microspheres SIRT | 3 months after treatment administration

SECONDARY OUTCOMES:
Progression Free Survival | Up to 12 months
Overall survival | Up to 30 months after inclusion of the 1st patient
Related Adverse Events in both arms as assessed by National Cancer Institute criteria (National Cancer Institute Common Terminology Criteria for Adverse Events, (NCI CTCAE) version 4). | Up to 12 months
Progression free survival not accessible to SIRT | Up to 12 months after treatment administration
Post-therapeutic dosimetry measured by Positron emission tomography-computed tomography PET / CT | Day one of treatment administration
  Dose delivered to the treated liver, the tumors, healthy liver and lings

CONTACTS AND LOCATIONS:
Overall Officials: Etienne GARIN, Pr, Study Chair — Centre Eugène Marquis
Locations (4):
- France (4):
  - CHU Henri Mondor, Créteil
  - CHU Saint Eloi, Montpellier
  - Centre Eugène Marquis, Rennes
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Garin E, Tselikas L, Guiu B, Chalaye J, Rolland Y, de Baere T, Assenat E, Tacher V, Palard X, Deandreis D, Mariano-Goulart D, Amaddeo G, Boudjema K, Hollebecque A, Meerun MA, Regnault H, Vibert E, Campillo-Gimenez B, Edeline J. Long-Term Overall Survival After Selective Internal Radiation Therapy for Locally Advanced Hepatocellular Carcinomas: Updated Analysis of DOSISPHERE-01 Trial. J Nucl Med. 2024 Feb 1;65(2):264-269. doi: 10.2967/jnumed.123.266211. PMID 38212068
- [Derived] Garin E, Tselikas L, Guiu B, Chalaye J, Edeline J, de Baere T, Assenat E, Tacher V, Robert C, Terroir-Cassou-Mounat M, Mariano-Goulart D, Amaddeo G, Palard X, Hollebecque A, Kafrouni M, Regnault H, Boudjema K, Grimaldi S, Fourcade M, Kobeiter H, Vibert E, Le Sourd S, Piron L, Sommacale D, Laffont S, Campillo-Gimenez B, Rolland Y; DOSISPHERE-01 Study Group. Personalised versus standard dosimetry approach of selective internal radiation therapy in patients with locally advanced hepatocellular carcinoma (DOSISPHERE-01): a randomised, multicentre, open-label phase 2 trial. Lancet Gastroenterol Hepatol. 2021 Jan;6(1):17-29. doi: 10.1016/S2468-1253(20)30290-9. Epub 2020 Nov 7. PMID 33166497